CLINICAL TRIAL: NCT06078150
Title: Effects of Active Video Games on Physical Activity, Mental Health, and Body Composition Among Overweight and Obese College Students in China
Brief Title: Effects of Active Video Games on Chinese Overweight and Obese College Students' Physical and Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Zhao Yue, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Zhao Yue
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Physical Inactivity; Mental Health Issue; Body Weight Changes
Keywords: Active Video Games; Overweight; Obesity; Physical Activity; Mental Health; Body Composition
MeSH Terms: conditions — Sedentary Behavior; Body Weight Changes; Overweight; Obesity; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The experimental group underwent a standardised AVG intervention according to the protocol of this experiment, and the control group did not do the intervention only recording daily life.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Active video game intervention for 1-6 weeks (Experimental): One hour three times a week for weeks 1-6 of the intervention (consisting of a 20-minute warm-up and a 40-minute AVG game).
  Interventions: Behavioral: Active video games intervention（1-6weeks）
- Experimental group: Active video game intervention for 7-12 weeks (Experimental): One hour three times a week for weeks 7-12 of the intervention (consisting of a 10-minute warm-up and a 50-minute AVG game).
  Interventions: Behavioral: Active video games intervention（7-12weeks）

INTERVENTIONS:
Behavioral: Active video games intervention（1-6weeks） — Experimental:
  Experimental group for weeks 1-3: enter the subject's basic information. The Fitness Ring Adventure requires subjects to be proficient in wearing two Joy-Con devices. Therefore, during the three interventions in the first week, subjects were able to fully understand how the AVG was worn, the game mechanics, and the game modes. Familiarise yourself with the warm-up and stretching patterns in the preparation phase of the game in order to be better prepared for subsequent interventions.
  Experimental group for weeks 4-6: to supervise and assist subjects during this intervention phase and to organize a speed passing competition at the end of week 6 to reward the subjects. Variables related to the subjects' activity, mental health, and physical composition were tested and recorded while testing proficiency in the game.
  Arms: Experimental group: Active video game intervention for 1-6 weeks
Behavioral: Active video games intervention（7-12weeks） — Experimental:
  Experimental group in weeks 7-9: continue to warm up before each game and then play the game. Passing tasks were set for each subject from week 7 onwards, and they had to pass 2 tasks during each weekly intervention.
  Experimental group in weeks 10-12: weekly intervention ensured that subjects were able to complete the pass 2 task, and if they completed the pass within the allotted time they were able to review the previously passed task. A boss fight was held in week 12, with a prize awarded to the person who took the shortest time.
  Arms: Experimental group: Active video game intervention for 7-12 weeks

SUMMARY:
Globally, overweight and obesity have become a major health concern and are present at all ages in both developed and developing countries. Sedentary lifestyle habits lead to reduced physical activity, which reduces energy expenditure, and this, combined with excessive energy intake, increases the risk of obesity. Lack of exercise combined with a sedentary lifestyle can exacerbate obesity and chronic disease. Among all obese people, the number of obese college students shows a growing trend. Obesity among college students not only leads to impaired physical health, but may also lead to discrimination, low self-confidence and self-efficacy, and even depression. Although traditional exercise methods can help college students with weight management, many college students do not enjoy these traditional physical activities. Therefore, there is an urgent need for a new form of exercise that is different from traditional exercise to get college students moving. Thus, obtaining the recommended level of physical activity.

With the progress of information technology and the popularity of electronic devices, the frequency of college students using computers and mobile phones has increased. Taking advantage of college students' interest in screen games, it is a new way to control sedentary behaviours and obesity by converting static screen usage time into dynamic screen usage time. Active video games (AVGs) are a new type of video games, which require players to complete the game by interacting with the images on the screen through upper limb, lower limb, and whole-body movements. Studies have shown that playing active video games produces more energy expenditure and physical activity than sedentary video games (static games).

The variety of research on AVGs is promising, but the population of participants in the studies has been mostly children and adolescents. The college student population, with a high prevalence of overweight and obesity, has a high prevalence of screen time. It is especially important to intervene with overweight and obese college students using AVG to shift their interest from screens to exercise, thereby increasing physical activity intensity. Therefore, this paper will systematically investigate the effects of AVGs on physical activity, mental health, and body composition of overweight and obese college students in China.

DETAILED DESCRIPTION:
To assess the effectiveness of AVG as an intervention modality, overweight and obese college students participating in this study are randomly assigned to two groups (experimental and control). The experimental group uses AVG as an intervention modality and the control group does not. Specifically, the experimental group uses Switch (OLED version), a Japanese console from Nintendo, with the game Fitness Ring Adventure for the intervention. The control group did not undergo the intervention and only followed their previous accustomed lifestyle in their daily lives. The total length of the experiment was 12 weeks and the intervention was conducted three times a week for one hour each time for the experimental group. The independent variable in this study was the AVG intervention; the dependent variables were physical activity, mental health, and body composition. Based on learning and summarising the research design of quantitative studies, the current study measured the dependent variable three times during the intervention period, including pre-test (pre-intervention), post-test1 (post-intervention week 6), and post-test2 (post-intervention week 12). The results of the three measurements of the dependent variable were collected, collated, and analyzed.

Physical activity is measured by calculating the number of steps using a pedometer (Yamax CW-700). Depression, stress, and anxiety were measured using the Depression Anxiety and Stress Scale (DASS) questionnaire, which consists of three self-reported scales designed to measure negative mood states such as depression, anxiety, and stress. Each of the three scales consists of 14 items with scores ranging from 0 to 42. The higher the total score, the greater the severity of the corresponding psychological problem. Previous studies have confirmed the validity of the depression, anxiety, and stress scales at 0.96, 0.89, and 0.93, respectively. Perceived need satisfaction was scored based on a revised 8-item statement using a 7-point Likert scale. Where 1 is (strongly disagree), 2 is (disagree), 3 is (fairly disagree), 4 is (unknown), 5 is (fairly agree), 6 is (agree), and 7 is (strongly agree). For example, "I felt camaraderie while playing this game", "I felt supported by the characters in the game" and "I really liked the characters I interacted with in this game". The scale has been validated with a Cronbach's alpha of 0.90. Subjects' enjoyment while participating in the experiment was measured using The Physical Activity Enjoyment Scale (PACES). The PACES is a 7-point scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) containing 16 declarative total scores ranging typically from 16 to 112, with higher scores indicating that the individual enjoys their physical activity The higher the score, the greater the enjoyment of the individual in physical activity. This scale has been validated in past studies and its Cronbach's alpha values were 0.88. Self-efficacy was measured by the Self-Efficacy Scale (GSES), which has 10 items and uses a 4-point Likert scale to measure the total score; the higher the score, the stronger the subject's self-efficacy. Exercise motivation was measured by Exercise Motivation Inventory-2 (EMI-2). The EMI-2 scale consists of 51 items, each of which is measured on a 6-point Likert scale ranging from 0 (not at all true for me) to 5 (very true for me), with higher scores indicating stronger exercise motivation. The variables to be measured for body composition were weight and body fat percentage. weight was measured using scales, BMI was calculated using a formula, body fat percentage was measured using bioelectrical impedance (BIA), and waist-to-hip ratio was measured using an accurate tape measure.

Before the training was conducted, all the people in the experimental group were explained, mainly including the registration of the account, the login of the game, and the explanation of the operation process. There are 23 levels in the game, each with different tasks and scenarios, requiring players to run, jump, and stretch to help the character reach the end and defeat the monsters for rewards. The experiment lasted 12 weeks, with three 1-hour interventions per week. For each intervention in weeks 1-6 of the experiment, a 20-minute warm-up (based on an animated cue before the official game) was performed, followed by 40 minutes of gameplay. For weeks 7-12 of the experiment, a 10-minute warm-up was performed followed by 50 minutes of gameplay.

Week 1: Firstly, register the Nintendo game account. After logging in, the origins of AVG games, and the gameplay and game modes of AVGs used in this experiment were introduced. Then the height, weight, and heart rate of the subjects were noted through the function that comes with the game. Then initially learned how to follow the virtual NPC on the TV screen for stretching operations and warm-up, and familiarised myself with the application and wearing of the fitness ring.

Week 2: Warm up according to the prompts of the game before each start. The warm-up included push and pull fitness rings, deep squats, stretching exercises, and free combination exercises. The warm-up time for each session was 20 minutes and the remaining 40 minutes were spent playing the game. The goal was set to two levels before each intervention. If the pass is completed you can continue to repeat the game for levels 1-2. In the second week subjects played levels 1-2.

Week 3: Followed the prompts of the AVG game to warm up and stretch before entering the formal game, this week performing levels 3-4.

Week 4: Follow the prompts of the AVG game for a warm-up and stretching then enter the formal game, play levels 5-6 this week.

Week 5: Follow the tips of the AVG game to warm up and stretch before moving on to the official game, playing levels 7-8 this week.

Week 6: Follow the tips of the AVG game to warm up and stretch before moving on to the official game, playing levels 9-10 this week. After the sixth week of testing, the first six weeks of play were reviewed and a speed play competition was held. Subjects were timed on how fast they could start 1-2 levels at a time. The shortest time was awarded.

Week 7: Follow the tips of the AVG game to warm up and stretch before moving on to the official game, playing levels 11-12 this week. From week 7 onwards, each intervention consisted of a 10-minute warm-up followed by 50 minutes of gameplay.

Week 8: Follow the tips of the AVG game for warm-up and stretching and then move on to the official game, playing levels 13-14 this week.

Week 9: Follow the tips of the AVG game to warm up and stretch and then move on to the official game, playing levels 15-16 this week.

Week 10: Follow the AVG game prompts to warm up and stretch before moving on to the official game, playing levels 17-18 this week.

Week 11: Follow the tips of the AVG game to warm up and stretch and then move on to the official game, playing levels 19-20 this week.

Week 12: Follow the tips of the AVG game to warm up and stretch before moving on to the official game, playing levels 21-23 this week. A review of all the games in the Fitness Ring Adventure. A competition in the monster-fighting mode is also held, requiring all subjects to defeat the monster of the difficult level in the shortest time. The person with the shortest time will receive a reward.

ELIGIBILITY:
Inclusion Criteria:

* Chinese university students between the ages of 18-22
* Overweight and obese Chinese university students (40≥BMI ≥ 25)
* No experience playing AVGs before participating in this experiment
* Subjects who were considered to be able to exercise healthily according to the Physical Activity Readiness Questionnaire (PAR-Q)
* There are no injuries to the ankle or upper or lower extremities that could affect participation in AVG intervention and daily life

Exclusion Criteria:

* College students majoring in physical education or involved in specialised training
* People who are pregnant or on a diet
* History of cardiorespiratory or respiratory disease (e.g., asthma) or metabolic disease
* Severe muscular or skeletal injuries within the past 3 months
* Participants with contraindications to physical activity as determined by the questions on the PAR-Q
* Other health problems that would affect the safety of the subject during the experiment.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Physical activity in overweight and obese university students | pretest, week 6, week 12
  Physical activity of overweight and obese college students was measured using a pedometer. The brand and model of the pedometer was the Yamax CW-700, and objective results of physical activity were obtained by measuring the number of steps with the pedometer, with more steps indicating greater physical activity.
Mental health of overweight and obese college students | pretest, week 6, week 12
  Depression, stress, and anxiety were measured using the Depression Anxiety and Stress Scale (DASS). There are a total of 42 questions, with scores ranging from 0 to 42. The higher the score, the greater the psychological problem. Perceived need satisfaction was scored on a revised 8-item statement using a 7-point Likert scale. High scores indicate high satisfaction with perceived needs. Enjoyment was measured using The Physical Activity Enjoyment Scale (PACES). PACES contains 16 statements with a score range of 16-112. Higher scores are more enjoyable. Self-efficiency was measured by the General Self-Efficiency Scale (GSES), which considerations of 10 items on a 4-point Likert scale. The higher the score, the stronger the self-efficiency of the participant. Exercise Motivation Inventory-2 (EMI-2) was used to measure motor motivation. The EMI 2 scale is composed of 51 items and each item is measured utilizing a 6-point Likert scale the higher scores indicate higher exercise motivation.
Body composition of overweight and obese college students | pretest, week 6, week 12
  Weight is measured using a standard kilogram scale and results are given in kilograms (kg), with weight accurate to 0.1kg.
  Body Mass Index (BMI) is measured using the formula BMI = weight (kg)/height (m)^2. Weight is expressed in kilograms and height in meters, with BMI being kg/m^2. Height is accurate to 0.1cm and weight is accurate to 0.1kg.
  Percentage of body fat was measured by a body composition analyzer using bioelectric impedance analysis (BIA), and the results were expressed in % (e.g., males with ≥25% body fat were considered obese; females with ≥30% body fat were considered obese).
  Waist-to-hip ratio was measured using an accurate tape measure, with waist and hip circumferences expressed in centimeters (cm) (e.g., waist-to-hip ratios greater than 0.9 for males and 0.85 for females were considered obese).

CONTACTS AND LOCATIONS:
Overall Officials: Yue Zhao, PhD, Principal Investigator — University Putra Malaysia
Locations (1):
- Qufu Normal University, Jining, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Result] Sousa CV, Hwang J, Cabrera-Perez R, Fernandez A, Misawa A, Newhook K, Lu AS. Active video games in fully immersive virtual reality elicit moderate-to-vigorous physical activity and improve cognitive performance in sedentary college students. J Sport Health Sci. 2022 Mar;11(2):164-171. doi: 10.1016/j.jshs.2021.05.002. Epub 2021 May 16. PMID 34004390
- [Result] Gao Z, Zeng N, McDonough DJ, Su X. A Systematic Review of Active Video Games on Youth's Body Composition and Physical Activity. Int J Sports Med. 2020 Aug;41(9):561-573. doi: 10.1055/a-1152-4959. Epub 2020 May 6. PMID 32375184
- [Result] Howe CA, Barr MW, Winner BC, Kimble JR, White JB. The physical activity energy cost of the latest active video games in young adults. J Phys Act Health. 2015 Feb;12(2):171-7. doi: 10.1123/jpah.2013-0023. Epub 2014 Jun 5. PMID 24905451
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/34004390/ — This article is from the National Library of Medicine.
- Available data/document: Systematic Review — https://pubmed.ncbi.nlm.nih.gov/32375184/ — This article is from the National Library of Medicine.
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/24905451/ — This article is from the National Library of Medicine.